CLINICAL TRIAL: NCT01859247
Title: Identification of Optimal Stimulation Site for Cervical Dystonia Symptoms: An Exploratory Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: Dystonia Coalition (Other); National Institutes of Health (NIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Sarah Pirio Richardson, MD, University of New Mexico
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: UNM 657; U54NS065701 (NIH)
Record Dates: First submitted 2013-05-09; First posted 2013-05-21 (Estimated); Results first posted 2016-07-28 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-06

CONDITIONS: Cervical Dystonia; Spasmodic Torticollis
Keywords: cervical dystonia; torticollis; rTMS
MeSH Terms: conditions — Torticollis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Dorsal Premotor rTMS (Active Comparator): 0.2 Hz rTMS for 15 minutes
  Interventions: Device: rTMS
- Primary motor cortex rTMS (Active Comparator): 0.2 Hz rTMS for 15 minutes
  Interventions: Device: rTMS
- Supplemental Motor Area rTMS (Active Comparator): 0.2 Hz rTMS for 15 minutes
  Interventions: Device: rTMS
- Anterior Cingulate rTMS (Active Comparator): 0.2 Hz rTMS for 15 minutes
  Interventions: Device: rTMS
- Sham rTMS (Sham Comparator): 0.2 Hz rTMS for 15 minutes
  Interventions: Device: rTMS

INTERVENTIONS:
Device: rTMS

SUMMARY:
The overall objective of this application is to therapeutically target the dysfunctional premotor-motor interaction in dystonia-and to provide a focused treatment of specific anatomical networks in order to reduce side effects and to improve symptom control over conventional therapies.

DETAILED DESCRIPTION:
We propose using repetitive transcranial magnetic stimulation (rTMS) over distinct premotor areas in patients with cervical dystonia (CD) with the goal of improving symptoms and reducing unwanted side effects. The knowledge gained in this proposed research will identify a specific premotor area to be targeted with rTMS that is expected to result in a novel intervention that could enhance or replace current treatments for CD. rTMS could be included as an adjunct treatment to botulinum toxin that could sustain treatment effect and decrease the frequency of re-injection, potentially resulting in cost savings without a decrease in symptom control. In addition to medical cost reduction, improved quality of life could be expected with the successful development of therapies that extend dystonia symptom control. rTMs has been FDA-approved for the treatment of depression and our proposal uses an even lower stimulation rate, suggesting continued use within clearly safe parameters. Successful completion of this research could lead to rapid adoption of this therapeutic modality.

We will test the hypothesis that rTMS of a distinct premotor site will provide more effective treatment of CD than non-specific activation of the entire premotor region. This will be done by performing a randomized, observer-blinded exploratory pilot study to determine the optimal site of rTMS over various sites of the premotor and motor cortex to improve the symptoms of cervical dystonia. Completion of this aim should lead to development of targeted TMS therapy for CD.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of idiopathic cervical dystonia
* Age 18 years or older
* Normal findings in the medical history, physical and neurological examination, except for dystonia
* Last treatment with botulinum toxin more than two months ago

Exclusion Criteria:

* History of seizure disorder
* Pregnancy- a pregnancy test will be performed for women of childbearing potential
* History of any other neurological disorders or conditions requiring the use of anti-depressants that are known to increase seizure threshold, neuroleptic medication, anticholinergic drugs and muscle relaxants
* History of neuroleptic medications/ prior use of neuroleptics

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-03; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Pirio Richardson, MD, Principal Investigator — University of New Mexico; H.A. Jinnah, MD, Study Director — Emory University
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

REFERENCES:
- [Background] Beck S, Houdayer E, Richardson SP, Hallett M. The role of inhibition from the left dorsal premotor cortex in right-sided focal hand dystonia. Brain Stimul. 2009 Oct;2(4):208-14. doi: 10.1016/j.brs.2009.03.004. Epub 2009 May 3. PMID 20633420
- [Background] Breakefield XO, Blood AJ, Li Y, Hallett M, Hanson PI, Standaert DG. The pathophysiological basis of dystonias. Nat Rev Neurosci. 2008 Mar;9(3):222-34. doi: 10.1038/nrn2337. PMID 18285800
- [Background] Lefaucheur JP, Fenelon G, Menard-Lefaucheur I, Wendling S, Nguyen JP. Low-frequency repetitive TMS of premotor cortex can reduce painful axial spasms in generalized secondary dystonia: a pilot study of three patients. Neurophysiol Clin. 2004 Oct;34(3-4):141-5. doi: 10.1016/j.neucli.2004.07.003. PMID 15501683
- [Background] Murase N, Rothwell JC, Kaji R, Urushihara R, Nakamura K, Murayama N, Igasaki T, Sakata-Igasaki M, Mima T, Ikeda A, Shibasaki H. Subthreshold low-frequency repetitive transcranial magnetic stimulation over the premotor cortex modulates writer's cramp. Brain. 2005 Jan;128(Pt 1):104-15. doi: 10.1093/brain/awh315. Epub 2004 Oct 13. PMID 15483042
- [Derived] Pirio Richardson S, Tinaz S, Chen R. Repetitive transcranial magnetic stimulation in cervical dystonia: effect of site and repetition in a randomized pilot trial. PLoS One. 2015 Apr 29;10(4):e0124937. doi: 10.1371/journal.pone.0124937. eCollection 2015. PMID 25923718

RESULTS

PARTICIPANT FLOW:
Groups:
- Subject 1: Received rTMS intervention in the following order, each at 0.2Hz for 15 minutes:
  Primary Motor Cortex Supplemental Motor Area Sham Dorsal Premotor Cortex Anterior Cingulate Cortex
- Subject 2: Received rTMS intervention in the following order, each at 0.2Hz for 15 minutes:
  Anterior Cingulate Cortex Primary Motor Cortex Dorsal Premotor Cortex Sham Supplemental Motor Area
- Subject 3: Received rTMS intervention in the following order, each at 0.2Hz for 15 minutes:
  Dorsal Premotor Cortex Supplemental Motor Area Sham Primary Motor Cortex Anterior Cingulate Cortex
- Subject 4: Received rTMS intervention in the following order, each at 0.2Hz for 15 minutes:
  Supplemental Motor Area Sham Anterior Cingulate Cortex Primary Motor Cortex Dorsal Premotor Cortex
- Subject 5: Received rTMS intervention in the following order, each at 0.2Hz for 15 minutes:
  Sham Dorsal Premotor Cortex Primary Motor Cortex Supplemental Motor Area Anterior Cingulate Cortex
- Subject 6: Received rTMS intervention in the following order, each at 0.2Hz for 15 minutes:
  Anterior Cingulate Cortex Dorsal Premotor Cortex Supplemental Motor Area Sham Primary Motor Cortex
- Subject 7: Received rTMS intervention in the following order, each at 0.2Hz for 15 minutes:
  Sham Primary Motor Cortex Dorsal Premotor Cortex Anterior Cingulate Cortex Supplemental Motor Area
- Subject 8: Received rTMS intervention in the following order, each at 0.2Hz for 15 minutes:
  Anterior Cingulate Cortex Supplemental Motor Area Primary Motor Cortex Sham Dorsal Premotor Cortex
Period: Overall Study
Arm/Group | Subject 1 | Subject 2 | Subject 3 | Subject 4 | Subject 5 | Subject 6 | Subject 7 | Subject 8
Started | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Completed | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Subject 1 | Subject 2 | Subject 3 | Subject 4 | Subject 5 | Subject 6 | Subject 7 | Subject 8 | Total
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 8
Age, Continuous [Mean (Full Range); unit: years] | 33 [33 to 33] | 60 [60 to 60] | 67 [67 to 67] | 31 [31 to 31] | 55 [55 to 55] | 41 [41 to 41] | 65 [65 to 65] | 72 [72 to 72] | 53 [31 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 3
  Male | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 8
TWSTRS Severity (Toronto Western Spasmodic Torticollis Rating Scale) [Mean (Full Range); unit: units on a scale] — Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) was used to assess severity of disease. The score for this section ranges from 0 (absence of severity) to 35 (maximum severity).
  units on a scale | 20 [20 to 20] | 9 [9 to 9] | 8 [8 to 8] | 14 [14 to 14] | 21 [21 to 21] | 20 [20 to 20] | 12 [12 to 12] | 16 [16 to 16] | 15 [8 to 20]
Dorsal Premotor-Motor Cortical Inhibition (DPMi) [Mean (Full Range); unit: Percentage] | 213 [213 to 213] | 127.50 [127.50 to 127.50] | 68.10 [68.10 to 68.10] | 71.60 [71.60 to 71.60] | NA [NA to NA] — Pre-DPMI not obtained | NA [NA to NA] — Pre-DPMI not obtained | 67.80 [67.80 to 67.80] | 72.30 [72.30 to 72.30] | NA [NA to NA] — Total not calculated because data are not available (NA) in one or more arms.
Cortical Silent Period (CSP) [Mean (Full Range); unit: milliseconds] | 169.10 [169.10 to 169.10] | 153.70 [153.70 to 153.70] | 133.28 [133.28 to 133.28] | 78.10 [78.10 to 78.10] | 136.92 [136.92 to 136.92] | 76.24 [76.24 to 76.24] | 113.16 [113.16 to 113.16] | 99.76 [99.76 to 99.76] | 105.03 [76.24 to 169.10]

OUTCOME MEASURES:

1. Primary Outcome: Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS)
Description: Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) was used to assess severity of disease. The score for this section ranges from 0 (absence of severity) to 35 (maximum severity).
Time Frame: Change from baseline pre-intervention TWSTRS score to post-intervention within 1 hour of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Primary Motor Cortex rTMS: 0.2Hz for 15 minutes
- Anterior Cingulate rTMS; Dorsal Premotor rTMS; Supplemental Motor Area rTMS; Sham rTMS: 0.2Hz for 15 minutes:
Arm/Group | Primary Motor Cortex rTMS | Anterior Cingulate rTMS | Dorsal Premotor rTMS | Supplemental Motor Area rTMS | Sham rTMS
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
units on a scale | -3.0 (4.8) | 0.25 (1.7) | -2.9 (3.4) | -1.5 (3.2) | -0.5 (1.1)

2. Secondary Outcome: Dorsal Premotor-motor Inhibition (dPMI)
Time Frame: Change from baseline dPMI to post-intervention within 1 hour of treatment
Population: two subjects did not have dPMI measured
Measure: Mean (Standard Deviation); unit: percentage
Groups:
- Anterior Cingulate rTMS; Dorsal Premotor rTMS; Supplemental Motor Area rTMS; Sham rTMS: 0.2Hz for 15 minutes
Arm/Group | Primary Motor Cortex rTMS | Anterior Cingulate rTMS | Dorsal Premotor rTMS | Supplemental Motor Area rTMS | Sham rTMS
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
percentage | 57.50 (40.5) | 2.10 (24.5) | 21.08 (42.5) | 32.21 (53.5) | 19.71 (80)

3. Secondary Outcome: Composite Measure of Patient Rating of Symptoms and Tolerability
Description: This measure will confirm the intervention tolerability by the patient. He/she scored the tolerability from 0-10, 0 being "completely tolerable" and 10 "completely intolerable."
Time Frame: Assessment completed immediately after rTMS treatment session
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Primary Motor Cortex rTMS | Anterior Cingulate rTMS | Dorsal Premotor rTMS | Supplemental Motor Area rTMS | Sham rTMS
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
units on a scale | 1.6 (1.8) | 1.6 (2.8) | 1.5 (2.7) | 0.9 (1.1) | 0.8 (1.0)

ADVERSE EVENTS:
Arm/Group | Subject 1 | Subject 2 | Subject 3 | Subject 4 | Subject 5 | Subject 6 | Subject 7 | Subject 8
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No